CLINICAL TRIAL: NCT03755609
Title: Efficacy of Oxycodone-propofol Combination Compared With a Fentanyl-propofol Combination on Conscious Sedation Effect and Early Cognitive Function During Therapeutic Endoscopic Retrograde Cholangio-pancreatography:a Prospective,Randomized, Single- Blinded Preliminary Trial
Brief Title: Efficacy of Oxycodone-propofol Combination Compared With a Fentanyl-propofol Combination on Conscious Sedation Effect and Early Cognitive Function During Therapeutic Endoscopic Retrograde Cholangio-pancreatography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Wuhan University (Other)
Responsible Party: Principal Investigator, fangjun, physician, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018006
Record Dates: First submitted 2018-11-16; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Conscious Sedation During Endoscopic Retrograde Choledochopancreatography
Keywords: Endoscopic Retrograde Choledochopancreatography; sedation; fentanyl; oxycodonel
MeSH Terms: interventions — Oxycodone; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients with oxycodone (Active Comparator)
  Interventions: Drug: Oxycodone
- patients with fentanyl (Sham Comparator)
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: Oxycodone — 0.1 mg/kg intravenously
  Arms: patients with oxycodone
Drug: fentanyl — 1ug/kg intravenously
  Arms: patients with fentanyl

SUMMARY:
To evaluate and compare the sedative effect and effects on early period cognitive function of a fentanyl-propofol Combination (FP) regimen with a oxycodone-propofol(OP) combination during the endoscopic retrograde cholangio-pancreatography (ERCP) requiring conscious sedation

DETAILED DESCRIPTION:
One hundred patients undergoing ERCP were included in this study and randomly divided into two groups of 50 people each. The patients in group FP were given fentanyl infusion of 1ug/kg intravenously 5 minutes before the process. They were given propofol infusion: a loading does of 1-2mg/kg immediately before the process then maintenance does of 1mg/kg/h. The patients in group OP were administered oxycodone of 0.1 mg/kg and 1-2mg/kg loading dose of propofol intravenously 5 minutes before the process. Then they were given 1mg/kg/h maintenance does of propofol infusion. In order to maintenan Ramsey Sedation Scale (RSS) between 3 and 4, all patients were administered 0.2~0.5 mg/kg bolus of propofol when necessary. Time of induction of anesthesia, operation time, wake-up time, recovery time, occurrence of adverse cardiovascular events, bucking, nausea and vomiting and respiratory depression ,total dosage of used propofol were assessed.Furthermore,different time point of regional cerebral oxygen saturation (rScO2) ,serum levels of irisin and cognitive function by mini-mental state examination (MMSE) were rated.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III

Exclusion Criteria:

* cardiovascular disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
anesthesia time | 2 days
operation time | 2 days

SECONDARY OUTCOMES:
irisin | 2 hours
  serum levels of irisin

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Guo P, Wu H, Liu L, Zhao Q, Jin Z. Efficacy of an Oxycodone-Propofol Combination versus a Fentanyl-Propofol Combination in Conscious Sedation during Therapeutic Endoscopic Retrograde Cholangiopancreatography in Elderly Patients. Gerontology. 2021;67(1):9-16. doi: 10.1159/000511173. Epub 2020 Dec 1. PMID 33260183